CLINICAL TRIAL: NCT00634075
Title: Clinical Assessment of Fish Oil-based Lipid Emulsion Infusions in Critical Patients With Severe Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Li Shin Hospital (Other)
Responsible Party: Boon-Siang Khor, Department of Emergency & Critical Care Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-08-01
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Severe Sepsis
Keywords: Severe sepsis; Proinflammatory cytokines; ICU
MeSH Terms: conditions — Sepsis | interventions — Docosahexaenoic Acids; fish oil triglycerides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: omega-3-fatty acids (Omegaven)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: omega-3-fatty acids (Omegaven) — The enrolled patients will be randomized to receive either supplementation of fish oil-based lipid emulsion (10 % Omegaven) as group 1 or placebo (0.9% Normal Saline) as group 2 via a central venous catheter within 24 hours after ICU admission, 100 ml daily for 5 days, respectively.
  Other Names: Omegaven
  Arms: 1
Drug: placebo — The enrolled patients will be randomized to receive either supplementation of fish oil-based lipid emulsion (10 % Omegaven) as group 1 or placebo (0.9% Normal Saline) as group 2 via a central venous catheter within 24 hours after ICU admission, 100 ml daily for 5 days, respectively.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a fish oil-based lipid emulsion, enriched with ω-3 fatty acids, reduce proinflammatory cytokines and mortality rate in critically ill patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Li Shin Hospital's ICU with a main diagnosis of severe sepsis.

Exclusion Criteria:

* Age of ﹤15 years
* Pregnancy
* Patients treated with immunosuppressive drugs or the equivalent of hydrocortisone more than 300 mg daily
* Plasma triglyceride concentration of more than 400 mg/dl
* Infection with human immunodeficiency virus
* Anticipated rapid fatality from irreversible underlying disease or malignancy
* Severe hemorrhagic disorders
* Acute myocardial infarction
* Recent stroke (within 3 month)
* Suspected or proven pulmonary embolism
* Cirrhotic liver and/or acute hepatitis ( elevation of serum GOT or GPT > 5 times of normal upper limit)
* Chronic renal failure (Cr >3.5 mg/dl upon admission) or end stage of renal diseases
* Allergic reactions against fish or egg proteins.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
All cause mortality | mortality rate on days 7 and 28.

SECONDARY OUTCOMES:
Lengths of ICU and hospital stay. Duration of mechanic ventilator requirement. Serial changing APACHE II and SOFA score. Changing of TNF-α, IL- 1β, IL-6, IL-8, and IL-10 levels. Incidence of hospital-acquired infection. | Days 0, 1, 3, 5, 7, 14 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Boon-Siang Khor, MD, Principal Investigator — Department of Emergency & Critical Care Medicine, Li Shin Hospital
Locations (1):
- Li Shin Hospital, Pingjen, Taoyuan County, Taiwan